CLINICAL TRIAL: NCT01761890
Title: Front-line Treatment of BCR-ABL+ Chronic Myeloid Leukemia (CML) With Dasatinib. An Observational Multicentric Study.
Brief Title: Front-line Treatment of BCR-ABL+ Chronic Myeloid Leukemia (CML) With Dasatinib
Acronym: CML1113
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CML1113; RSO ID 714 (Other: Observational Study Register)
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; Early phase; CML; Dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CML patients
  Interventions: Behavioral: Dasatinib discontinuation

INTERVENTIONS:
Behavioral: Dasatinib discontinuation — Treatment decision is at the discretion of the investigator and must not be made on the basis of this observational study. Patients should have their treatment initiated in accordance with the summary of product characteristics.

SUMMARY:
The GIMEMA CML Working Party promotes a multicentric, observational, non company sponsored, prospective study of Chronic Myeloid Leukemia (CML) patients treated frontline with dasatinib. Patients will be followed for 5 years. This study will help the definition of guidelines for the treatment of CML patients in early phases.

The primary objective of the study is to describe, in the clinical practice, the rate of events leading to permanent discontinuation after 2 years of treatment with dasatinib as frontline therapy in newly diagnosed CML patients.

DETAILED DESCRIPTION:
The primary objective is to describe, in the clinical practice, the rate of events leading to permanent discontinuation after 2 years of treatment with dasatinib as frontline therapy in newly diagnosed CML patients. Imatinib mesylate, a protein tyrosine kinase inhibitor (TKI) targeting BCR-ABL, has become in the last decade the standard of care for Chronic Myeloid Leukaemia (CML) in chronic phase (CP)1-3. Dasatinib is a second generation TKI, effective in imatinib-resistant and imatinib-intolerant patients, which demonstrated superior efficacy to imatinib in early CP BCR-ABL+ CML patients 4,6,7. Most data on second generation TKIs are from company-sponsored studies, generally implemented in selected referral centres. The long-term outcome is still unknown. The high rate of study discontinuation observed within the phase 3 study may influence the mid-term and the long-term data interpretation6,7. A long-term post-marketing surveillance in large independent trial is extremely important to confirm the feasibility of a frontline treatment with the second generation TKI dasatinib and to evaluate the efficacy in a nationwide experience. Moreover, obtaining a deep molecular response is extremely relevant in order to consider TKIs discontinuation. This condition is known as "Complete Molecular Response" (CMR) and is further defined according to the sensitivity achieved (for the definition see the "Criteria of evaluation" section). As far as treatment discontinuation, two experiences have been published so far, aimed at evaluating the persistence of the CMR after imatinib discontinuation. The first was a pilot study32 where 12 patients were included. These 12 patients discontinued imatinib after at least 2 years of CMR (median duration of negativity, 32 months). Six patients displayed a molecular relapse with a detectable BCR-ABL transcript at 1, 2, 3, 4, and 5 months. Imatinib was then reintroduced and led to a novel molecular response. Six other patients (50%) still have an undetectable level of BCR-ABL transcript after a median follow-up of 18 months (range, 9-24 months). The results of this pilot trial have been confirmed and extended in a second trial, the STIM trial33: 100 patients were enrolled, median follow-up 17 months, 69 patients with at least 12 months follow-up: 42 (61%) of these 69 patients relapsed (40 before 6 months, one patient at month 7, and one at month 19). At 12 months, the probability of persistent CMR for these 69 patients was 41% (95% CI 29-52). All patients who relapsed responded to reintroduction of imatinib. An increase of the CMR rate could possibly translate in a higher proportion of patients candidate to stopping anti-CML treatment, with higher probability of remaining disease-free in the long term. Interestingly, dasatinib was able to induce higher 36-month cumulative MR4 and MR4.5 rates than imatinib7. The advantages of this possible future scenario could be: first, the possibility of treatment discontinuation at least in patients with chronic clinical adverse events; second, a potential reduction of the costs of TKI treatment (after the introduction of TKI, the costs of CML treatment is increasing year by year, with the increasing prevalence of CML patients).

In summary, 1) Most data on second generation TKIs are from company-sponsored studies; 2) The high rate of study discontinuation observed within the phase III study may influence the data interpretation; 3) A long-term post-marketing surveillance in large independent trial is extremely important to confirm the efficacy in a nationwide experience; 4) The persistence of CMR after TKI discontinuation have been described in selected patients with "deep" molecular response; 5) A stable CMR is a pre-requisite for treatment discontinuation; 6) A detailed description of the kinetic of the molecular response, potentially related to a subsequent treatment discontinuation, will be done.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetic and/or molecular confirmed diagnosis of Ph+ and/or BCR-ABL+ CML; Age 18 years;
* Early chronic phase, less than 6 months from diagnosis. Prior treatment with Hydroxyurea or Anagrelide is allowed;
* Signed written informed consent according to ICH/EU/GCP and national local laws prior to any study procedures.

Exclusion Criteria:

* Prior treatment with any protein tyrosin-kinase inhibitor (TKI) or interferon;
* Recommendations and precautions before allocating a new CML case to dasatinib are fully described in the prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicentre, observational, prospective study of newly diagnosed chronic phase CML patients treated frontline with Dasatinib 100 mg QD.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of dasatinib permanent discontinuing patients. | After 2 years from study entry.
  The cumulative rate of dasatinib permanent discontinuation by 2 years.

SECONDARY OUTCOMES:
Number of dasatinib permanent discontinuing patients. | After 5 years from study entry.
  The cumulative rate of dasatinib permanent discontinuation by 5 years.
Number of confirmed MR4 and MR4.5. | After 2 years from study entry.
  The rate of confirmed MR4 and MR4.5 by 24 months.
Number of confirmed MR4 and MR4.5. | After 60 months from study entry.
  The rate of confirmed MR4 and MR4.5 by 60 months.
Number of stable MR4 and MR4.5 and characteristics. | After 60 months from study entry.
  The stability of MR4 and MR4.5.
Number of Complete Cytogenetic Responses (CCgR) | After one year from study entry.
  The rate of Complete Cytogenetic Response (CCgR) at 1 year.
Number of Major Molecular Response (MMR). | After one year from study entry.
  The rate of Major Molecular Response (MMR) at 1 year.
Number of days to response (CCgR, MMR, MR4, MR4.5). | After 4 years from study entry.
  The median time to response and the overall estimated probability of response (CCgR, MMR, MR4, MR4.5).
Number of overal surviving patients | After five years from study entry.
Number of progression-free survival patients. | After five years from study entry.
Number of failure-free survival patients. | After five years from study entry.
Number of event-free survival patients. | After five years from study entry.
Number of responses | After 7 years from study entry.
  Overall responses and long-term outcome according to baseline prognostic factors (including: Sokal score34, Euro score35 and EUTOS score36; presence of additional chromosomal abnormalities in Ph+ cells; BCR-ABL transcript type; comorbidity score index).
Number of responses according to BCR-ABL transcript levels. | After 3 and 6 months from study entry.
  Overall responses and long-term outcome according to BCR-ABL transcript levels and CgR at 3 months and at 6 months.
Number of patients with fasting glucose modifications. | After 24 months from study entry.
  Fasting glucose modifications (diabetic and normo-glycemic patients) and HbA1C modifications (diabetic patients only) during the first 24 months.
Number of patients with modifications of body mass index during treatment compared to baseline. | After 7 years from study entry.
  Modifications of body mass index during treatment compared to baseline.
Number of patients with modifications of serum lipids during treatment compared to baseline. | After 7 years from study entry.
  Modifications of serum lipids during treatment compared to baseline.
Patient reported quality of life. | At 3, 6, 9, 12, 18, 24 months from study entry.
Number of adverse events. | At 3, 6, 9, 12, 18, 24 months from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, Pr., Study Chair — Orsola Malpighi, Bologna
Locations (37):
- Italy (37):
  - Centro Oncologico Basilicata, Rionero in Vulture, Potenza
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - US Dipartimentale - Centro per le malattie del sangue - Ospedale Civile - S.Giacomo, Castelfranco Veneto
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Ferrara
  - Azienda Ospedaliera di Firenze, Florence
  - Centro Aziendale di Ematologia ASL N. 6, Livorno
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - zienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - zienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Rotondo Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation — http://www.gimema.it